CLINICAL TRIAL: NCT06273761
Title: Primary Care Community Pharmacy Project: Evaluation of Medication Management Service
Brief Title: Evaluation of Medication Management Service
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other); Hong Kong Sheng Kung Hui Welfare Council Limited (Other); Hong Kong Young Women's Christian Association (Other); Haven of Hope Hospital (Other); Pok Oi Hospital (Other); St. James' Settlement (Other); Aberdeen Kai-fong Welfare Association (Other); Health In Action (Unknown); Lok Sin Tong Benevolent Society, Kowloon (Other)
Responsible Party: Principal Investigator, Prof. Ian Chi Kei Wong, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW 23-550
Record Dates: First submitted 2024-01-09; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-01

CONDITIONS: Medication Adherence; Medication Safety; Diabetes Mellitus, Type 2; Hypertension; Polypharmacy; High Risk Medications
Keywords: Medication Management Service; Community pharmacy service
MeSH Terms: conditions — Medication Adherence; Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants who join the trial will have have a control period (no intervention) of 3 to 12 months before receiving medication management service (MMS) at 8 NGO community pharmacies. Since there are 8 NGO community pharmacies, 2 NGO community pharmacies will start delivering MMS by phase at 3, 6, 9 and 12 month intervals. Therefore, all participants who join the trial will receive MMS by month 12 from recruitment date. During the MMS service, pharmacists will review the participants' medication history and conduct medication reconciliation, refer them to doctors for reviewing the prescribing decision if necessary, as well as provide education and lifestyle advice on medication management.
  Interventions: Behavioral: Medication Management Service (MMS)
- Control (No Intervention): Participants who join the trial will have have a control period of 3 to 12 months before receiving medication management service (MMS) at 8 NGO community pharmacies. Participants will have no MMS intervention during the control period. Since there are 8 NGO community pharmacies, two NGO community pharmacies will start delivering MMS by phase at 3, 6, 9 and 12 month intervals. Therefore, all participants who join the trial will receive MMS by month 12 from recruitment date.

INTERVENTIONS:
Behavioral: Medication Management Service (MMS) — Medication Management Service (MMS) is a service delivered by community pharmacists aiming at helping patients resolve their medication therapy problems (MTPs) by carrying out medication reconciliation, provision of education about their medication regimen, and also providing professional pharmacological advice to patients.
  Arms: Intervention

SUMMARY:
Medication management services (MMS) is a pharmacist-led service of optimizing the medication use and health outcomes, by promoting medication safety and enhancing the ability in self-management of health and diseases of patients and their caregivers. Yet, only limited evidence on the implementation of MMS service in Hong Kong is available. The goal of this clinical trial is to evaluate the cost effectiveness and effects of implementing MMS in community pharmacies owned by 8 non-government organizations (NGOs) in Hong Kong on humanistic and clinical outcomes in patients with hypertension and/or type II diabetes mellitus. The clinical trial aims to look into the following aspects:

* To evaluate the perception and satisfaction of patients on MMS service
* To investigate whether MMS could improve patients' adherence to their medication regimen, health-related quality of life, health outcomes and health service utilization, as well as their ability to understand and cope with their illness and drug-related problems
* To identify and categorize the types of drug-related problems identified during MMS
* To evaluate the cost-effectiveness of implementing MMS in community pharmacies

MMS services will be rolled out in a total of 8 NGO community pharmacies progressively (2 pharmacies per phase) in 4 successive phases. Participants will complete the questionnaires at the following time points throughout the trial, namely 1) during recruitment, 2) baseline (1 month before MMS), 3) 3 months after MMS begins, 4) 12 months after MMS begins, and 5) 24 months after MMS begins. Researchers will compare the results of questionnaires conducted at different time points to identify the potential changes in the effects of MMS. Furthermore, researchers will link up the electronic health records of the participants and identify the potential changes in the health outcomes and health service utilizations after receiving MMS.

DETAILED DESCRIPTION:
This is a randomized controlled trial which will be conducted across 8 NGO community pharmacies in Hong Kong. The order of providing MMS service by 8 NGO community pharmacies to study participants will be determined by randomization. The time before each NGO community pharmacy provides MMS service to the study participants is considered as the control period (no MMS service will be provided). A total of 8 NGO community pharmacies will be divided into 4 groups and hence 2 pharmacies will have the same length of control period. The control periods will be categorized into 3-month, 6-month, 9-month and 12-month long. It is anticipated that a total of 640 participants will be recruited to the trial. Informed written consent will be obtained from the study participants before the study starts. Since this trial will involve accessing to personal and healthcare information of study participants for analysis, informed written consent will also be sought for the authorization to access clinical data on the Electronic Health Record Sharing System (eHealth) and the electronic health records from the Hospital Authority (HA) for service evaluation and research purposes. Eligible participants will receive MMS service provided by the pharmacists who work in the NGO community pharmacies after the control period. Different study instruments and methods will be used to evaluate humanistic, clinical and economic outcomes.

To evaluate the humanistic outcomes, participants will complete the validated questionnaires at 5 different time points throughout the trial, namely 1) during recruitment, 2) baseline (1 month before MMS), 3) 3 months after MMS begins, 4) 12 months after MMS begins, and 5) 24 months after MMS begins. Descriptive statistics will be conducted to summarize the participants' characteristics and outcomes of interest. Linear and nonlinear mixed effect models will be conducted for continuous and binary outcomes, respectively.

To evaluate the clinical outcomes, electronic health records of the trial participants will be extracted from the electronic health database of the HA. The HA is the statutory organization that coordinates all public hospitals and primary care clinics, and is responsible for managing the majority of patients with chronic diseases in Hong Kong. Participants' demographics, medical records and clinical parameters will be collected from the HA clinical management system database. Clinical parameters such as blood pressure and blood glucose level will be used to evaluate the differences between before and after MMS. In addition, the attendance and admission records of A&E and hospitalization will also be collected to evaluate the changes in the health service utilization before and after MMS.

For the evaluation of economic outcomes, a costing study will be conducted to collect the set-up costs and operation costs of MMS service via sending questionnaires to the 8 NGO community pharmacies. Participants will complete the validated questionnaire on health-related quality of life (EQ-5D) to estimate quality-adjusted life years (QALYs). The differences in health service utilization, medical costs and QALYs in participants before and after using MMS will be estimated. The Incremental cost-effectiveness ratio (ICER) based on incremental cost per additional QALY would be calculated. Probabilistic sensitivity analysis based on Monte Carlo simulation will be conducted to test the robustness of estimated costs and QALYs. Finally, a cost-effectiveness acceptability curve will be constructed to assess the simulated probability over a range of amounts that a decision-maker might be willing to pay the MMS for an additional QALY.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* diagnosed with Type 2 diabetes mellitus and/or hypertension
* having regular follow-up on Type 2 diabetes mellitus and/or hypertension at Hospital Authority
* no A&E admission/hospitalization in the past 3 months
* no recent changes in medication regimen in the past 3 months
* polypharmacy (taking 5 or more chronic medications)
* using at least 1 high-risk medication (Anticoagulants, Oral hypoglycaemics, Insulins, psychotropic medications or immunosuppressants)
* able to communicate in Cantonese and/or English

Exclusion Criteria:

* aged below 18
* unable to give informed consent
* unable to communicate in Cantonese and/or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | Medication adherence will be assessed at 5 time points, namely 1) during recruitment, 2) baseline (1 month before MMS), 3) 3 months after MMS begins, 4) 12 months after MMS begins, and 5) 24 months after MMS begins.
  Medication adherence will be assessed by the Medication Adherence Report Scale (MARS-5) which consists of a total of 5 items and is used to assess patient's adherence to their medications. Participants rate items on a 5-point scale. The score range for MARS-5 is 5-25, higher score indicates better adherence to take medications.

SECONDARY OUTCOMES:
Additional health service utilization | Through study completion, an average of 1 year
  Changes in health service utilization (e.g. A&E admission, hospitalization) before and after receiving medication management service will be assessed using record linkage to the electronic health records from the Hospital Authority.
Patient perception and satisfaction | Patient perception and satisfaction will be assessed at 3 time points, namely 1) 3 months after MMS begins, 2) 12 months after MMS begins, and 3) 24 months after MMS begins.
  Patient perception and satisfaction will be assessed by the Pharmacy Services Questionnaire (PSQ). The PSQ consists of 20 items and will be rated by participants on a 5-point scale. (5-Excellent, 4- Very good, 3-Good, 2-Fair and 1-Poor). The maximum score is 100 and the minimum score is 20. Higher scores indicate high levels of satisfaction.
Patient perceived sensitivity to medicines | Patient perceived sensitivity to medicines will be assessed at 3 time points, namely 1) 3 months after MMS begins, 2) 12 months after MMS begins, and 3) 24 months after MMS begins.
  Perceived Sensitivity to Medicines Scale (PSM-5) will be used to assess the patient's perception on their sensitivity to medicines. Patients will rate the items on a 5-point scale. (5-Strongly agree, 4- Agree, 3-Neutral, 2-Disagree and 1-Strongly disagree).The maximum score is 25 and the minimum score is 5. Higher scores indicate stronger perceived sensitivity to medicines.
Social impact | Social impact will be assessed at 5 time points, namely 1) during recruitment, 2) baseline (1 month before MMS), 3) 3 months after MMS begins, 4) 12 months after MMS begins, and 5) 24 months after MMS begins.
  Social impact will be assessed by the Patient Enablement Index (PEI). The PEI is a 6-item questionnaire and is used to assess patient enablement. The maximum score of PEI is 12 and minimum score is 0. Higher scores indicate greater levels of enablement and a score of 0 indicates no enablement.
Health-related quality of life | Health-related quality of life will be assessed at 5 time points, namely 1) during recruitment, 2) baseline (1 month before MMS), 3) 3 months after MMS begins, 4) 12 months after MMS begins, and 5) 24 months after MMS begins.
  Health-related quality of life will be assessed by the EuroQol EQ-5D-5L (EQ-5D-5L). The EQ-5D-5L is a 5-item questionnaire used to assess health-related quality of life. The maximum score of EQ-5D-5L is 25 and the minimum score is 5. Higher scores indicate better health status. EQ-5D visual analog scale records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher health related quality of life.
Drug-related problems | Throughout the study period, up to 24 months.
  The number of drug-related problems will be extracted from the computerized clinical documentations system input by the pharmacists.
Change in costs | Throughout the study period, up to 24 months.
  A costing questionnaire will be used for extracting set-up and operational costs of delivering Medication Management Services. Change in health service utilization rate will be obtained from the electronic health records managed by Hospital Authority (HA). Cost associated with the health service utilization will be obtained from the HA Gazette. Change in costs is defined by the difference between before and after MMS intervention.
Change in effectiveness | Throughout the study period, up to 24 months.
  Effectiveness will be measured by quality adjusted life years (QALYs), which will be derived from the EQ-5D-5L adjustment weights. Change in effectiveness is defined by the difference between before and after MMS intervention.
Incremental cost effectiveness ratio (ICER) | Throughout the study period, up to 24 months.
  Incremental cost effectiveness ratio (ICER) is defined as changes in cost divided by changes in QALYs.
Beliefs in medicines | Beliefs in medicines will be assessed at 5 time points, namely 1) during recruitment, 2) baseline (1 month before MMS), 3) 3 months after MMS begins, 4) 12 months after MMS begins, and 5) 24 months after MMS begins.
  The Beliefs about Medicines Questionnaire (BMQ) is a 23-item questionnaire used to assess medication beliefs and perceptions toward medications. The BMQ consists of BMQ-General and BMQ-Specific. BMQ-General is used to assess beliefs that medicines are overused (General-Overuse), medicines are harmful (General-Harm) and medicines are beneficial (General-Benefit). BMQ-Specific assesses beliefs about the necessity of medicines to maintain health (Specific-Necessity) and concerns about potential adverse effects of medicines (Specific-Concerns). Items are scored on a 5-point Likert scale. The score range for BMQ is 23-115. Higher scores indicate stronger beliefs in the subscale.

CONTACTS AND LOCATIONS:
Locations (8):
- Hong Kong (8):
  - Aberdeen Kai-Fong Welfare Association A-Lively Community Pharmacy, Hong Kong
  - Health In Action Community Pharmacy, Hong Kong
  - Hong Kong Sheng Kung Hui Welfare Council Community Pharmacy, Hong Kong
  - PHARM+ Haven of Hope Community Pharmacy, Hong Kong
  - PHARM+ Pok Oi Hospital Community Pharmacy, Hong Kong
  - PHARM+ St. James' Settlement Community Pharmacy, Hong Kong
  - PHARM+ The Lok Sin Tong Community Pharmacy, Hong Kong
  - PHARM+ YWCA Community Pharmacy, Hong Kong

IPD SHARING:
Plan to Share IPD: No